CLINICAL TRIAL: NCT05833724
Title: A Phase II, Open-label, Single-arm, Multicenter Study of Chidamide in Patients With Relapsed or Refractory Peripheral T-cell Lymphoma
Brief Title: Chidamide in Patients With Relapsed or Refractory Peripheral T-cell Lymphoma (R/R PTCL)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Great Novel Therapeutics Biotech & Medicals Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KEPIDA-2
Record Dates: First submitted 2023-04-17; First posted 2023-04-27 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2024-12

CONDITIONS: Relapsed or Refractory Peripheral T-cell Lymphoma
Keywords: PTCL
MeSH Terms: conditions — Recurrence; Lymphoma, T-Cell, Peripheral | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; HBI-8000

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chidamide (Experimental): Chidamide tablets orally, twice a week.
  Interventions: Drug: Chidamide

INTERVENTIONS:
Drug: Chidamide — Subjects will receive a single dose of 30 mg chidamide. Twice a week.
  Other Names: Tucidinostat; HBI-8000

SUMMARY:
This is a phase II, open-label, non-randomized, single-arm, multicenter study to evaluate the efficacy, safety, and PK of chidamide in patients with R/R PTCL.

DETAILED DESCRIPTION:
This is a phase II, open-label, non-randomized, single-arm, multicenter study to evaluate the efficacy, safety, and PK of chidamide in patients with R/R PTCL. To determine eligibility, subjects must have PTCL confirmed with a sample or specimen evaluated by the investigator.A treatment cycle is defined as 4 weeks. All eligible subjects will be treated with chidamide until disease progression, intolerable toxicity effects, death, or withdrawal of consent.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathological diagnosis, made by the investigator, of the following PTCL subtypes as defined by the WHO classification (2016) may be included: PTCL, not otherwise specified (PTCL-NOS), anaplastic lymphoma kinase-positive (ALK+) anaplastic large-cell lymphoma (ALCL), ALK-negative (ALK-) ALCL, angioimmunoblastic T-cell lymphoma (AITL), extranodal natural killer (NK)/T-cell lymphoma, nasal type (ENKL), etc., except cutaneous form or leukemic form.
2. Patients for whom at least one measurable lesion according to Cheson Criteria 2014 at baseline.
3. Relapsed or refractory disease (including DOR shorter than 30 days) to ≥1 prior systemic therapy including, but not limited to, chemotherapy, target therapy, immunotherapy, and autologous stem cell transplantation.
4. Male or female, aged 20-75 years (inclusive).
5. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
6. With a life expectancy of ≥12 weeks.
7. Have not received radiotherapy, chemotherapy, immunotherapy (except for antibody therapy), or target therapy within 4 weeks prior to the start of study drug.
8. Have not received any antibody therapy within 12 weeks prior to the start of study drug.
9. Willing to provide written informed consent.

Exclusion Criteria:

1. Females who are pregnant or breastfeeding, or females of childbearing potential who are not willing to use adequate contraception.
2. Patients in whom central nervous system lymphoma is recognized during screening (if suspected clinically, imaging study should be performed to confirm).
3. Have been treated with histone deacetylase (HDAC) inhibitor.
4. With a history of clinically significant QTc prolongation (>450 ms for males or >470 ms for females), ventricular tachycardia (VT), atrial fibrillation (AF), heart block (HB), myocardial infarction (MI) onset within one year, congestive heart failure (CHF), or any other symptomatic coronary artery disease requiring treatment.
5. The size of fluid area detected by cardiac ultrasonography in cavum pericardium is ≥10 mm during diastolic period.
6. With a history of organ transplantation.
7. With a history of allogeneic stem cell transplantation.
8. Have received autologous stem cell transplantation within 12 weeks prior to the start of study drug.
9. Have participated in a clinical trial involving investigational antibody therapy within 12 weeks prior to the start of study drug or non-antibody therapy within 4 weeks prior to the start of study drug.
10. Have received symptomatic treatment for early myelotoxicity within 7 days prior to the start of study drug.
11. With active bleeding or newly diagnosed thromboembolic disease, or with hemorrhagic tendency who are using anticoagulants.
12. With active infection of hepatitis B or C, or persistent fever within 14 days prior to the start of study drug.
13. With history of testing positive for human immunodeficiency virus or known acquired immunodeficiency syndrome.
14. Had a major organ surgery within 6 weeks prior to the start of study drug.
15. With abnormal hepatic function (serum total bilirubin >1.5 x upper limit of normal [ULN]; alanine aminotransferase [ALT]/aspartate aminotransferase [AST] >2.5 x ULN or >5 x ULN if liver metastases are present), abnormal renal function (serum creatinine >1.5 x ULN), or abnormal complete blood count (absolute neutrophil counts <1500/μL; platelet counts <90 x 1000/μL, hemoglobin <9 g/dL).
16. Has known psychiatric disorders or substance abuse disorders that may interfere with the patient's participation in the study or evaluation of the study results.
17. Considered by the investigator as being not suitable to participate the study.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2024-10-18 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 24 months
  Objective response rate was defined as the percentage of participants with a complete response (CR) or a partial response (PR) according to International Working Group (IWG) criteria. The response was assessed based on clinical and radiological criteria. CR is defined as the disappearance of all evidence of disease. PR is defined as a regression of measurable disease and no new sites. As pre-defined, the primary endpoint analysis for this study was based on the Independent Overall Efficacy Review Committee (IOERC) assessment of response.

SECONDARY OUTCOMES:
Time to response (TTR) | 24 months
  Time to response was defined as the time (in weeks) from first administration of treatment until first response. Response is defined as complete response (CR) or partial response (PR). CR is defined as the disappearance of all evidence of disease. PR is defined as a regression of measurable disease and no new sites.
Duration of response (DOR) | 24 months
  The Duration of Response was assessed by IWG criteria per the IRC from the date the measurement criteria were first met for CR or PR (whichever status was recorded first) until the first subsequent date that relapse or progression was documented. Response is defined as complete response (CR) or partial response (PR). CR is defined as the disappearance of all evidence of disease. PR is defined as a regression of measurable disease and no new sites.
Progression-free survival (PFS) | 24 months
  Progression-free survival (PFS) was the duration of time from first administration of study treatment to date of first documented progression or death from any cause. It was based on tumor assessments made according to the IWG criteria as assessed by the IRC. The progression is defined as any new lesion or increase by ≥ 50% of previously involved sites from nadir.
Overall survival (OS) | 24 months
  Overall Survival was the time from first administration of study treatment until the date of death.
Pharmacokinetics profiles - (AUC0-t) | Blood samples collected on Days 1-4 and 25-28 of Cycle 1, pre-dose and up to 72 hours post-dose (28 days/cycle)
  Area under the plasma concentration-time curve from time zero to time t(AUC0-t)
Pharmacokinetics profiles - (AUC0-∞) | Blood samples collected on Days 1-4 and 25-28 of Cycle 1, pre-dose and up to 72 hours post-dose (28 days/cycle)
  Area under the plasma concentration-time curve from time zero to infinity(AUC0-∞)
Pharmacokinetics profiles - (Cmax) | Blood samples collected on Days 1-4 and 25-28 of Cycle 1, pre-dose and up to 72 hours post-dose (28 days/cycle)
  Maximum plasma concentration(Cmax)
Pharmacokinetics profiles - (Tmax) | Blood samples collected on Days 1-4 and 25-28 of Cycle 1, pre-dose and up to 72 hours post-dose (28 days/cycle)
  Time to maximum plasma concentration(Tmax)
Pharmacokinetics profiles - (T1/2) | Blood samples collected on Days 1-4 and 25-28 of Cycle 1, pre-dose and up to 72 hours post-dose (28 days/cycle)
  Half-life(T1/2)
Pharmacokinetics profiles - (Ctrough) | PK samples collected on Day 15, Day 18, and Day 22 predose (28 days/cycle)
  Pre-dose trough concentration (Ctrough)

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Nan Chen, Ph.D., Study Director — Great Novel Therapeutics Biotech & Medicals Corporation
Locations (5):
- Taiwan (5):
  - Chang Gung Memorial Hospital, Kaohsiung, Kaohsiung City
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Chang Gung Memorial Hospital, Linkou, Taoyuan District

IPD SHARING:
Plan to Share IPD: Undecided